CLINICAL TRIAL: NCT01848847
Title: The Impact of Bladder Distention on Execution of Diagnostic Hysteroscopy Procedure; a Randomised Controlled Trial.
Brief Title: Relationship Between Bladder Distention and Hysteroscopy Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, CEM CELIK, Assistant Professor, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 9598
Record Dates: First submitted 2013-04-10; First posted 2013-05-08 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-07

CONDITIONS: Menorrhagia
Keywords: Hysteroscopy; Bladder; Pain; Feasibility; Duration
MeSH Terms: conditions — Menorrhagia; Pain | interventions — Hysteroscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full Bladder (Experimental): Hysteroscopy conducted under full bladder.
  Interventions: Procedure: Hysteroscopy
- Empty Bladder (Experimental): Hysteroscopy conducted under empty bladder.
  Interventions: Procedure: Hysteroscopy

INTERVENTIONS:
Procedure: Hysteroscopy

SUMMARY:
The purpose of the study is to investigate the advantages and disadvantages of bladder filling during hysteroscopy procedure.

DETAILED DESCRIPTION:
Women who should have diagnostic hysteroscopy procedure will be randomly allocated into two groups. In the first group hysteroscopy will be performed with a filled bladder and in the second group procedure will be performed with an empty bladder. The women will be assigned into groups randomly. The duration of the procedure, feasibility of the procedure and tolerability of procedure will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Women who are at reproductive age
* Women who are not pregnant at the time of presentation
* Women who are not nulliparous

Exclusion Criteria:

* Women who have previous cervical surgery or cervical incompetence.
* Women who have genitourinary infection
* Women who have profuse uterine bleeding or recent uterine perforation
* Women who have neurological disorders affecting evaluation of pain.

Ages: 17 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cem Celik, Assist Prof, Study Director — Namik Kemal University Faculty of Medicine Department of Obstetrics and Gynecology
Locations (1):
- Namık Kemal University Faculty of Medicine Department of Obstetric and Gynecology, Tekirdağ, Turkey (Türkiye)

REFERENCES:
- [Background] Kabli N, Tulandi T. A randomized trial of outpatient hysteroscopy with and without intrauterine anesthesia. J Minim Invasive Gynecol. 2008 May-Jun;15(3):308-10. doi: 10.1016/j.jmig.2008.01.013. Epub 2008 Mar 20. PMID 18439502
- [Background] Carta G, Palermo P, Marinangeli F, Piroli A, Necozione S, De Lellis V, Patacchiola F. Waiting time and pain during office hysteroscopy. J Minim Invasive Gynecol. 2012 May-Jun;19(3):360-4. doi: 10.1016/j.jmig.2012.01.017. Epub 2012 Mar 3. PMID 22387163
- [Background] De Iaco P, Marabini A, Stefanetti M, Del Vecchio C, Bovicelli L. Acceptability and pain of outpatient hysteroscopy. J Am Assoc Gynecol Laparosc. 2000 Feb;7(1):71-5. doi: 10.1016/s1074-3804(00)80012-2. PMID 10648742
- [Background] Pansky M, Feingold M, Bahar R, Neeman O, Asiag O, Herman A, Sagiv R. Improved patient compliance using pediatric cystoscope during office hysteroscopy. J Am Assoc Gynecol Laparosc. 2004 May;11(2):262-4. doi: 10.1016/s1074-3804(05)60211-3. PMID 15200787

RESULTS

PARTICIPANT FLOW:
Groups:
- Empty Bladder: Hysteroscopy conducted under empty bladder.
  Hysteroscopy : bladder filling before diagnostic outpatient hysteroscopy
- Full Bladder: Hysteroscopy conducted under full bladder.
  Hysteroscopy : bladder filling before diagnostic outpatient hysteroscopy
Period: Overall Study
Arm/Group | Empty Bladder | Full Bladder
Started | 51 | 51
Completed | 49 | 48
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Empty Bladder | Full Bladder | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 48 | 97
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.51 (7.04) | 41.07 (7.68) | 40.27 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 48 | 97
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 49 | 48 | 97

OUTCOME MEASURES:

1. Primary Outcome: Ease of Cervical Entry
Description: Ease of cervical entry which will be assessed by Likert scale.The outcome measures in this study were the ease of cervical entry (judged by the individual surgeons using a 5-point Likert scale: very difficult= 1, difficult= 2, fair = 3, easy= 4, and very easy = 5.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Empty Bladder | Full Bladder
Number analyzed (Participants) | 49 | 48
units on a scale | 4.00 (0.86) | 3.55 (0.90)

2. Secondary Outcome: Patient Acceptability and Pain Scoring
Description: Patient acceptability and pain scoring will be evaluated by Likert scale and visual analog scale.
Time Frame: two months
Reporting Status: Not Posted

3. Secondary Outcome: Procedure Duration
Description: Procedural time which will be measured in minutes
Time Frame: two months
Reporting Status: Not Posted

4. Primary Outcome: Pain Scoring(VAS)
Description: Pain scoring was made by 10 cm visual analog scale. pain score (recorded by the patient on a 10 -point visual analog scale (VAS) which means pain increases with increasing number
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Empty Bladder | Full Bladder
Number analyzed (Participants) | 49 | 48
units on a scale | 2.52 (1.2) | 1.95 (1.1)

ADVERSE EVENTS:
Arm/Group | Empty Bladder | Full Bladder
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/47
Other Adverse Events (participants affected / at risk) | 0/49 | 0/47

LIMITATIONS AND CAVEATS:
difficulties in introduction of hysteroscopy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes